CLINICAL TRIAL: NCT03735017
Title: Immersive Virtual Walking Treatment for Neuropathic Pain in Spinal Cord Injury
Brief Title: Virtual Reality Walking for Neuropathic Pain in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Zina Trost, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 383546
Record Dates: First submitted 2018-10-31; First posted 2018-11-08 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain
Keywords: Virtual Reality
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two intervention arms. Both groups receive the same number of sessions, duration of sessions, and measures procured.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and key research staff assessing outcomes will be blind to condition allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Interactive (Active Comparator): Participants will receive non-interactive virtual reality walking sessions.
  Interventions: Other: Non-Interactive Virtual Reality Walking
- Interactive (Experimental): Participants will receive interactive virtual reality walking sessions.
  Interventions: Other: Interactive Virtual Reality Walking

INTERVENTIONS:
Other: Non-Interactive Virtual Reality Walking — Individuals will wear a head-mounted display to allow them to visualize virtual legs in the virtual environment. When wearing the display, individuals will see the legs and arms of their virtual avatar from a first-person perspective.
  Individuals will engage in virtual reality sessions in their home twice daily over the course of 10 days in a two-week period. Each daily session will take approximately 30 minutes, with 5-10 minutes dedicated to the virtual walking experience. Additionally, each daily session will be scheduled a minimum of 4 hours apart.
  Arms: Non-Interactive
Other: Interactive Virtual Reality Walking — Individuals will wear a head-mounted display to allow them to visualize virtual legs in the virtual environment. When wearing the display, individuals will see the legs and arms of their virtual avatar from a first-person perspective.
  Individuals will engage in virtual reality sessions in their home twice daily over the course of 10 days in a two-week period. Each daily session will take approximately 30 minutes, with 5-10 minutes dedicated to the virtual walking experience. Additionally, each daily session will be scheduled a minimum of 4 hours apart.
  Arms: Interactive

SUMMARY:
This study will examine the effectiveness of one of two virtual reality treatments on neuropathic pain in individuals with spinal cord injury.

DETAILED DESCRIPTION:
The investigators are investigating the effectiveness of one of two possible investigational virtual reality treatments on neuropathic pain in individuals with spinal cord injury. Participants will be randomized to one of these two treatments.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with complete paraplegic spinal cord injury who report chronic neuropathic pain
* Individuals with persistent spinal cord injury neuropathic pain
* More than one - year post injury
* Stable medication regimen for the past month

Exclusion Criteria:

* Conditions that impair movement of the arms
* Significant cognitive impairment as suggested by apparent incomprehension of screening questions as judged by the evaluator
* For those for whom voluntary arm movement would cause sufficient discomfort (>4/10) that could prevent trial completion will be excluded from participation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-06-16 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Pain Intensity as assessed by Numeric Rating Scale | Baseline - Final assessment (average 1 week post treatment)
  The Numeric Rating Scale (NRS) measures pain intensity measured via 0-10 numeric rating scale.
  Range of scores: 0-10
Neuropathic Pain Qualities as assessed by Neuropathic Pain Scale | Baseline - Final assessment (average 1 week post treatment)
  The Neuropathic Pain Scale (NPS) was designed to assess the distinct pain qualities associated with neuropathic pain.The NPS consists of 10 items. Seven of the 10 items contain the words intense, sharp, hot, dull, cold, and itchy to characterize the patient's pain and the word sensitive to describe the patient's pain reaction to light touch or clothing.One item describes the time quality of the pain (all the time or some of the time). The ninth item describes the overall unpleasantness of the pain, whereas the last item indicates the intensity of the deep and surface pain. In the NPS each item is rated separately. All the items are rated 0-10 scale, with higher score indicative of more neuropathic pain for each type of respective pain.
  Range of scores: 0-10 for each item.
Neuropathic Pain Diagnosis as assessed by Doleur Neuropatique 4 | Baseline - Final assessment (average 1 week post treatment)
  Doleur Neuropatique 4 is a 10 item survey that evaluates neuropathic pain following central and neurological lesions. It has components of how the pain feels to the patient (e.g. burning, cold, electrical shocks, tingling, hypoaesthesia). Responses to each item is yes or no, with each yes response equaling one point.
  Range of scores: 0-10. 4/10 and greater indicate neuropathic pain.
Pain Interference specific to spinal cord injury as assessed by International Spinal Cord Injury Pain Basic Data Set version 2.0 | Baseline - Final assessment (average 1 week post treatment)
  Pain interference measured International Spinal Cord Injury Pain Basic Data Set version 2.0 interference items. There are 3 pain interference items using a 0-10 numeric rating scale for each item. Items can be assessed by summing the score or by individual assessment of items.
  Summed range of scores: 0-30. Individual item range of scores: 0-10
Pain Interference as assessed by Brief Pain Inventory | Baseline - Final assessment (average 1 week post treatment)
  Pain interference measured by Brief Pain Inventory interference items. 7 items each use a 0-10 scale. Item scores may be assessed individually, or by taking the average score of all items.
  Range of Scores: 0-10. Increased scores indicate higher levels of interference due to pain.

SECONDARY OUTCOMES:
Patient Treatment Evaluation as assessed by the Ease of Usefulness, Satisfaction, and Ease of Use Questionnaire | Final assessment (average 1 week post treatment)
  Ease of Usefulness, Satisfaction, and Ease of use Questionnaire is a 30 item survey. Subscales include: treatment's usefulness, ease of use, ease of learning, and satisfaction. Each item is presented on a 7-point Likert scale. Each subscale is calculated by averaging all items in subscale.
  Range of scores for each subscale: 1-7
Patient Treatment Evaluation as assessed by the Patient Global Impression of Change Scale | Final assessment (average 1 week post treatment)
  Patient treatment evaluation is assessed by the Patient Global Impression of Change. This is a one item 7 point Likert item assessing improvement of the participants overall status.
  Range of scores: 1-7
Patient Treatment Evaluation as assessed by the Modified Treatment Evaluation Inventory | Final assessment (average 1 week post treatment)
  Patient treatment evaluation is assessed by Treatment Evaluation Inventory. This is a 9 item scale with a 5-point Likert responses for each question. The items are scored by summing all items.
  Range of scores: 9-45. A higher score indicates greater acceptance of treatment.
Patient Treatment Evaluation as assessed by Semi-structured Qualitative Interviewing | Final assessment (average 1 week post treatment)
  Patient treatment evaluation is assessed by semi-structured interviewing. Qualitative feedback from participant experience will be assessed by thematic analyses.
Quality of Life and Participation are assessed by the SF-36 Walk-Wheel | Baseline - Final assessment (average 1 week post treatment)
  Quality of life and participation are assessed by the SF-Walk Wheel. This is a 36 item assess health concepts which represent basic human values and were relevant to a person's functional status and well-being. The responses are based on a Likert scale. There are the following subscales: Physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health.
  Each item is recoded to a preset value between 0-100 per the scoring key.
  Range of scores: 0-100 for each sub-scale. A higher score defines a more favorable health state.
Quality of Life is assessed by Satisfaction with Life Scale | Baseline - Final assessment (average 1 week post treatment)
  Quality of life is assessed by the Satisfaction with Life Scale. This is a 5 item survey. Response options are a 7-point Likert scale. Items may be assessed individually or by summing items.
  Range of scores: 5-35. Higher scores indicate more satisfaction in life
Depression and mood are assessed by the Patient Health Questionnaire -9 | Baseline - Final assessment (average 1 week post treatment)
  Depression and mood are measured by Patient Health Questionnaire-9. This is a 10 item tool. The first 9 items are a 4-point Likert scale assessing depressive symptoms. The first 9 items are summed to determine depressive symptom severity. Item 10 assesses difficulty dealing with items 1-9. Item 10 is not used in scoring severity.
  Range of scores: 0-27. Higher scores indicate more depressive symptom severity.
Perceived Disability is assessed by the Pain Disability Index | Baseline - Final assessment (average 1 week post treatment)
  Perceived Disability measured by a modified Pain Disability Index. The rating scales are designed to measure the degree to which aspects of life are disrupted by chronic pain. This is a 7 item survey with response options of 0-10. Each item may be assessed individually, or by summing all items.
  Individual item range of scores: 0-10 Total range of scores: 0-70. The higher the index, the greater the person's disability due to pain.
Absorption is assessed by the Tellegen Absorption Scale | Baseline
  Tellegen Absorption Scale is a 34-item multi-dimensional measure that assesses imaginative involvement and the tendency to become mentally absorbed in everyday activities. Item responses are on a 5-point Likert scale. Items are summed to score.
  Range of scores: 0-136. Higher scores indicate greater levels of absorption.
Immersive Tendencies are assessed by the Immersive Tendencies Questionnaire | Baseline
  Immersive Tendencies are assessed by the Immersive Tendencies Questionnaire (ITQ). This is an 18-item survey. Item responses use a 7 point Likert scale. Subscales include: focus, involvement, emotions, and play. Each subscale is scored by summing items. A total score is scored by summing all items.
  Range of total score: 18-126 Focus range of scores: 5-35 Involvement range of scores: 5-35 Emotions range of scores: 4-28 Play range of scores: 3-21 Higher scores indicate higher immersive tendencies overall and in each sub-scale.
fMRI Imaging | Baseline - Final assessment (average 1 week post treatment)
  We are studying pain by functional Magnetic Resonance Imaging (fMRI) which allows us to identify certain parts of the brain that show how the brain works in controlling pain perception and cognitions.

CONTACTS AND LOCATIONS:
Overall Officials: Zina Trost, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Trost Z, Anam M, Seward J, Shum C, Rumble D, Sturgeon J, Mark V, Chen Y, Mitchell L, Cowan R, Perera R, Richardson E, Richards S, Gustin S. Immersive interactive virtual walking reduces neuropathic pain in spinal cord injury: findings from a preliminary investigation of feasibility and clinical efficacy. Pain. 2022 Feb 1;163(2):350-361. doi: 10.1097/j.pain.0000000000002348. PMID 34407034